CLINICAL TRIAL: NCT02359305
Title: Institutional Audit of the Use of Intravenous Acetaminophen in Infants Undergoing Pyloromyotomy
Status: Completed | Type: Observational
Sponsor: Arlyne Thung (Other)
Responsible Party: Sponsor-Investigator, Arlyne Thung, Clinical Assistant Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB14-00149
Record Dates: First submitted 2014-07-31; First posted 2015-02-10 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-04

CONDITIONS: Pyloric Stenosis
MeSH Terms: conditions — Pyloric Stenosis | interventions — Acetaminophen

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- IV Acetaminophen: Acetaminophen administered by intravenous infusion.
  Interventions: Drug: Acetaminophen
- Rectal Acetaminophen: Acetaminophen administered by rectal suppository.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen given by IV
  Other Names: Ofirmev
  Groups: IV Acetaminophen
Drug: Acetaminophen — Acetaminophen suppository given rectally
  Other Names: Acephen, Feverall
  Groups: Rectal Acetaminophen

SUMMARY:
This is a retrospective chart review. The objective of the current study is to determine the analgesic efficacy and side effect profile of intravenous acetaminophen when administered to infants undergoing pyloromyotomy. In addition, recovery characteristics of infants who were administered intravenous acetaminophen will be compared to infants who did not receive intravenous acetaminophen to determine if there were any appreciable differences with regard to postoperative discomfort, PACU time, time to oral feeds and hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* patients who presented for pyloromyotomy

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who presented for pyloromyotomy
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Acetaminophen: Acetaminophen given by intravenous infusion.
- Rectal Acetaminophen: Acetaminophen given by rectal suppository.
Period: Overall Study
Arm/Group | IV Acetaminophen | Rectal Acetaminophen
Started | 34 | 34
Completed | 34 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen | Rectal Acetaminophen | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34 | 34 | 68
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 34.2 (14.5) | 37.8 (16.5) | 36 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 29 | 29 | 58
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 68

OUTCOME MEASURES:

1. Primary Outcome: Acetaminophen Dosage
Description: One time in the OR prior to the start of surgery
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | IV Acetaminophen | Rectal Acetaminophen
Number analyzed (Participants) | 34 | 34
mg/kg | 8.6 (3.9) | 30.7 (6.3)

2. Primary Outcome: Average FLACC Pain Score in the PACU
Description: The Face, Legs, Activity, Cry, Consolability scale or FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain.
Time Frame: 0-60 minutes post-operatively
Measure: Mean (Standard Deviation); unit: units on a scale 0-10
Arm/Group | IV Acetaminophen | Rectal Acetaminophen
Number analyzed (Participants) | 34 | 34
units on a scale 0-10 | 0.3 (0.6) | 0.6 (1)

3. Secondary Outcome: PACU Time
Description: Time spent in the post-anesthesia care unit post-operatively.
Time Frame: 45-60 minutes post-operatively
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | IV Acetaminophen | Rectal Acetaminophen
Number analyzed (Participants) | 34 | 34
minutes | 48 (19.9) | 50.4 (12)

ADVERSE EVENTS:
Time Frame: During hospital stay following surgery (average 1-3 days).
Arm/Group | IV Acetaminophen | Rectal Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes